CLINICAL TRIAL: NCT04912232
Title: Continued Development of a Multiplex Precision Medicine System for Early Warning of Progression Toward Hemodynamic Deterioration After Trauma
Brief Title: Trauma Study: Early Warning of Progression Toward Hemodynamic Deterioration After Trauma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant funding for the study ended.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Dartmouth College (Other); Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY02001495
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2023-06

CONDITIONS: Occult Bleeding; Hemorrhage
Keywords: Occult Bleeding; Hemorrhage; Hemorrhagic Shock; Trauma Injury; Precision Medicine; Triage; Bioimpedance; Electrical Impedance Tomography; Electrical Impedance Spectroscopy; Near-Infrared Spectroscopy
MeSH Terms: conditions — Hemorrhage; Shock, Hemorrhagic; Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Trauma Patients (Experimental): Patients suffering blunt and/or penetrating trauma but without physiologic criteria suggestive of ongoing hemorrhage:
  1. Awake and alert GCS >14
  2. Admission systolic blood pressure greater than 90 and heart rate less than 120
  3. Without signs of clinically significant ongoing external hemorrhage with no active bleeding documented on radiology/ultrasound and stable vital signs (no signs of hemodynamic deterioration) during initial evaluation (approximately 15 minutes post admission)
  Interventions: Device: Detection of Occult Hemorrhage in Trauma Patients

INTERVENTIONS:
Device: Detection of Occult Hemorrhage in Trauma Patients — Non-invasive monitoring of trauma patients

SUMMARY:
This study is Phase 3 of a three-phase DOD CDMRP funded project for the development of a multi-technology poly-anatomic noninvasive system for early detection of occult hemorrhage.

Early detection of ongoing hemorrhage (OH) before onset of shock is a universally acknowledged great unmet need, and particularly important after trauma. Delays in the detection of OH are associated with a "failure to rescue" and a dramatic deterioration in prognosis once the onset of clinically frank shock has occurred. An early alert to the presence of OH with an acceptable rate of false-positives and false-negatives would save countless lives. Additionally, such technology would save significant time, money and effort by allowing medical resources to be applied more accurately - the essence of precision medicine. An automated system would monitor currently stable patients continuously, leaving clinicians free to care for patients in need of attention.

DETAILED DESCRIPTION:
The investigators will enroll 480 trauma patients in a "no significant risk" prospective clinical trial to 1) evaluate the performance of a Mark I prototype, 2) validate the performance of the Phase II algorithm, and 3) re-train the algorithm to Phase III iteration.

This is not a therapeutic study. The main outcome variables are non-invasive measurements that will be used for machine learning, not real-time patient management. The data generated will be used later for discovery and validation in traditional and innovative machine learning.

As a minimal risk study, there will be no change from standard of care for patients undergoing surgery. The surgical procedures and pharmacotherapies will proceed as per standard clinical management.

Enrolled patients will undergo standard preoperative, anesthetic, and postoperative physiological monitoring that includes:

Electrocardiogram: Heart rate and electrical activity of the heart will be recorded via a 3-lead ECG.

Arterial Oxygen Saturation (SpO2): Pulse oximetry will be recorded using a commercially available finger pulse oximeter.

Finger Photoplethysmography: waveforms will be obtained non-invasively from either the SpO2 photoplethysmography or alternatively a Flashback Technologies Compensatory Reserve Index (CRI™) device.

In addition to these standard physiologic measurements, as a part of the research, the investigators will also acquire the following non-invasive optical and impedance measurements. All of these devices have been previously validated as non-invasive and safe in humans. The impedance electrodes and optical emitter/detectors will be incorporated into easily applied latex-free based "belts" that will be applied to anatomic locations along the thorax, abdomen and thigh. Application of these belts will be as soon as practical after patient arrival.

The clinicians providing care to the patient will be blind with respect to the measurements from these devices.

Continuous-wave Near-Infrared Spectroscopy (CW-NIRS) Device, custom built:

The device is built on an Ocean Optics FLAME USB Spectrometers, with two OSRAM 4736 NIR LEDs in plastic holders meant to be taped or strapped to the patient on the chest/torso and thigh locations. An Oceans Optics tungsten-halogen light source is used for an additional probe location on the forehead. Probe holders are designed to collect light from surface of skin by means of a mirror and collimator. The device will collect data on light attenuation of muscle in models of shock/trauma. The light output for all locations is below the ANSI limits for maximum permissible skin exposure.

SwissTom Electrical Impedance Tomography (EIT) System:

Name of device: Pioneer Set (Electrical Impedance Tomography System) Device Manufacturer: SwissTom AG (Parent company SenTec AG)

This device monitors dynamically changing perfusion physiology. To record multiplexed impedance signature a belt of 16-32 electrodes is placed around the thorax above the nipple line and thigh and impedances are recorded between multiple sets of electrodes.

SwissTom develops a clinical EIT system that is approved for pulmonary imaging. This Pioneer system is their research platform that has similar functionality and safety performance to their clinical system but provides research teams with access to raw data and additional functionality for specifying imaging parameters (e.g. control of frame rates, signal frequency acquisition, electrode drive patterns).

ScioSpec MultiChannel Electrical Impedance Spectroscopy (EIS) System:

Name of device: ISX-Mini (MultiChannel Electrical Impedance Spectroscopy System) Device Manufacturer: ScioSpec

To record multiplexed impedance signatures- an array of 4 electrodes is placed around the cranium and thorax of the patient and impedance spectroscopy signatures are recorded at each anatomic location. This device monitors dynamically changing intracranial, intrathoracic and intra-abdominal physiology.

General Approach to Minimize Risk:

This protocol will be minimal risk to patients as there is little risk associated with the placement of these devices and they can be removed at any time. They don't interfere with standard equipment used in clinical management of trauma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Awake and alert GCS >14
2. Admission systolic blood pressure greater than 90 and heart rate less than 120
3. Without signs of clinically significant ongoing external hemorrhage with no active bleeding documented on radiology/ultrasound and stable vital signs (no signs of hemodynamic deterioration) during initial evaluation (approximately 15 minutes post admission)

Exclusion Criteria:

1. Altered mental status GCS < 13
2. Systolic blood pressure less than 90 or heart rate greater than 120
3. Need for ongoing fluid or pressor support (standard local fluid resuscitation only)
4. Clinically significant ongoing external hemorrhage
5. Respiratory distress with O2 saturation <96%
6. Pre-existing systemic illness, likely to alter systemic cardiovascular response to hemorrhage (overt clinical heart failure). Including congestive heart failure, and a paced cardiac rhythm.
7. Pregnant
8. Prisoner status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noman Paradis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share IPD.

REFERENCES:
- [Background] Shackelford SA, Colton K, Stansbury LG, Galvagno SM Jr, Anazodo AN, DuBose JJ, Hess JR, Mackenzie CF. Early identification of uncontrolled hemorrhage after trauma: current status and future direction. J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 2):S222-7. doi: 10.1097/TA.0000000000000198. No abstract available. PMID 24770559
- [Background] Parks JK, Elliott AC, Gentilello LM, Shafi S. Systemic hypotension is a late marker of shock after trauma: a validation study of Advanced Trauma Life Support principles in a large national sample. Am J Surg. 2006 Dec;192(6):727-31. doi: 10.1016/j.amjsurg.2006.08.034. PMID 17161083
- [Background] Wo CC, Shoemaker WC, Appel PL, Bishop MH, Kram HB, Hardin E. Unreliability of blood pressure and heart rate to evaluate cardiac output in emergency resuscitation and critical illness. Crit Care Med. 1993 Feb;21(2):218-23. doi: 10.1097/00003246-199302000-00012. PMID 8428472
- [Background] Convertino VA, Moulton SL, Grudic GZ, Rickards CA, Hinojosa-Laborde C, Gerhardt RT, Blackbourne LH, Ryan KL. Use of advanced machine-learning techniques for noninvasive monitoring of hemorrhage. J Trauma. 2011 Jul;71(1 Suppl):S25-32. doi: 10.1097/TA.0b013e3182211601. PMID 21795890
- [Background] Convertino VA. Blood pressure measurement for accurate assessment of patient status in emergency medical settings. Aviat Space Environ Med. 2012 Jun;83(6):614-9. doi: 10.3357/asem.3204.2012. PMID 22764618
- [Background] Kim SH, Lilot M, Sidhu KS, Rinehart J, Yu Z, Canales C, Cannesson M. Accuracy and precision of continuous noninvasive arterial pressure monitoring compared with invasive arterial pressure: a systematic review and meta-analysis. Anesthesiology. 2014 May;120(5):1080-97. doi: 10.1097/ALN.0000000000000226. PMID 24637618
- [Background] Soller BR, Yang Y, Soyemi OO, Ryan KL, Rickards CA, Walz JM, Heard SO, Convertino VA. Noninvasively determined muscle oxygen saturation is an early indicator of central hypovolemia in humans. J Appl Physiol (1985). 2008 Feb;104(2):475-81. doi: 10.1152/japplphysiol.00600.2007. Epub 2007 Nov 15. PMID 18006869
- [Background] Belle A, Ansari S, Spadafore M, Convertino VA, Ward KR, Derksen H, Najarian K. A Signal Processing Approach for Detection of Hemodynamic Instability before Decompensation. PLoS One. 2016 Feb 12;11(2):e0148544. doi: 10.1371/journal.pone.0148544. eCollection 2016. PMID 26871715

RESULTS

PARTICIPANT FLOW:
Groups:
- Trauma Patients: Patients suffering blunt and/or penetrating trauma but without physiologic criteria suggestive of ongoing hemorrhage:
  1. Awake and alert GCS >14
  2. Admission systolic blood pressure greater than 90 and heart rate less than 120
  3. Without signs of clinically significant ongoing external hemorrhage with no active bleeding documented on radiology/ultrasound and stable vital signs (no signs of hemodynamic deterioration) during initial evaluation (approximately 15 minutes post admission)
  Detection of Occult Hemorrhage in Trauma Patients: Non-invasive monitoring of trauma patients
Period: Overall Study
Arm/Group | Trauma Patients
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Algorithm Performance: Time of Alarm Before Onset of Deterioration
Time Frame: patient data will be collected over 3-6 hours
Population: Only 1 participant was enrolled was stable for 6 hours (no signs of hemodynamic deterioration). Therefore there was no data to analyze algorithm performance. Algorithm developed was to be trained to alarm under two circumstances indicating significant risk of ongoing hemorrhage progressing to shock: 1) a change from baseline, 2) development of prespecified patterns. This participant did not experience a triggering event, and therefore there was no data to be used to evaluate the algorithm.
Measure: Number; unit: minutes
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
minutes | NA — lack of events

2. Primary Outcome: Algorithm Performance: Sensitivity as Measured by for Alarm/no Alarm Outcome
Time Frame: patient data will be collected over 3-6 hours
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
percent | NA — Lack of events

3. Primary Outcome: Algorithm Performance: Specificity as Measured by for Alarm/no Alarm Outcome
Time Frame: patient data will be collected over 3-6 hours
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
percent | NA — lack of events

4. Primary Outcome: Algorithm Performance: Positive Predictive Value for Alarm/no Alarm Outcome
Time Frame: patient data will be collected over 3-6 hours
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
percent | NA — lack of events

5. Primary Outcome: Algorithm Performance: Negative Predictive Value for Alarm/no Alarm Outcome
Time Frame: patient data will be collected over 3-6 hours
Population: as for outcome 1
Measure: Number; unit: percent
Arm/Group | Trauma Patients
Number analyzed (Participants) | 1
percent | NA — lack of events

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Trauma Patients
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT04912232/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT04912232/ICF_001.pdf